CLINICAL TRIAL: NCT06919978
Title: Effect of Position to Prevent Pleural Irritation (PPPI) on Pain Level and Sleep Quality in Patients With Chest Tube: A Single-blind Quasi-experimental Study.
Brief Title: Position to Prevent Pleural Irritation (PPPI) for Pain and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Emine Kol, Professor, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSA-2018-3765
Record Dates: First submitted 2025-02-01; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chest Tube; Thoracotomy; Pain; Sleep
Keywords: Thoracic surgery; Pleural irritation; Chest tube irritation; Sleep quality; Pain control; Positioning in bed
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: The study was conducted in a non-randomized, single-blind, quasi-experimental design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Position to Prevent Pleural Irritation (PPPI) Group (Experimental): The participants in the Position to Prevent Pleural Irritation (PPPI) group were positioned in bed in order to minimize pleural irritation caused by the contact of the chest tube with the pleura during sleep.
  Interventions: Behavioral: The Position to Prevent Pleural Irritation (PPPI)
- Routine care (No Intervention): Participants in the control group received routine care in the clinical procedure. Participants assumed their desired in-bed position for sleep.

INTERVENTIONS:
Behavioral: The Position to Prevent Pleural Irritation (PPPI) — The Position to Prevent Pleural Irritation (PPPI) was administered once before sleep on the first night of the day the participant arrived at the clinic.
  Arms: The Position to Prevent Pleural Irritation (PPPI) Group

SUMMARY:
Clinical Trial Aim: The study was conducted to investigate the effect of the Position given to Prevent Pleural Irritation (PPPI) due to chest tube on pain level and sleep quality in patients undergoing thoracic surgery.

Does the Position to Prevent Pleural Irritation (PPPI) reduce participants' pain levels due to pleural irritation? Does the Position to Prevent Pleural Irritation (PPPI) improve participants' sleep quality? Researchers were compare the effectiveness of the Position to Prevent Pleural Irritation (PPPI) in reducing pain from pleural irritation and improving sleep quality with routine clinical care.

Participants received the in-bed position and the Position to Prevent Pleural Irritation (PPPI) applied by the researcher in routine care before their first night's sleep in the clinic after thoracotomy. At the same time, participants' pain was be assessed with a pain scale, and their sleep quality was be assessed with a PolySomnioGraph (PSG) and sleep scale.

DETAILED DESCRIPTION:
The participants in the study group were positioned in bed the Position to Prevent Pleural Irritation (PPPI) in order to minimize pleural irritation caused by the contact of the chest tube with the pleura during sleep. Routine care was applied by the researcher in the clinic's prosedure for the participants in the control group.

Position to Prevent Pleural Irritation (PPPI)

1. The participants were informed before the surgery and consent was obtained. The positioning and sleep measurement method were explained. Sleeping scale was filled out for information about the sleep routine before hospitalization.
2. When the participants were admitted to the thoracic surgery clinic, information about positioning and sleep measurement was given by the researcher.
3. The researcher questioned and evaluated the patient's pain before bedtime, and routine analgesic were applied.
4. It was checked that the participant's bed was in working order for the Position to Prevent Pleural Irritation (PPPI), and the positions that could be given with the bed's remote control were explained to the participant.
5. The position and working order of the chest drainage system and drainage tube were checked.
6. The participant was given an upright or dorsal recumbent position with the head of the bed at 30-45 degrees, according to participant's preference. Pillows were placed under the head, under the shoulder where the tube was located, and under the arms, according to the participant's preference. In order to keep the abdominal muscles relaxed, femur and knee flexion was provided.
7. PolySomnioGraph (PSG) was placed on the participant for sleep measurement. The participant's satisfaction about the position was questioned. The room lights were turned off, and noise-causing factors were removed.
8. In the morning, the PolySomnnioGraph (PSG) connections were removed from the participant and pain was questioned and rated again.

ELIGIBILITY:
Inclusion Criteria:

* being in the 18-70 age group (adult age group accepted for pain perception and sleep)
* being operated on by the same surgical team
* having a posterolateral thoracotomy technique
* having the same anesthesia and analgesia protocol
* being transferred from the intensive care unit to the clinic at the 48th hour after thoracotomy
* having a single chest tube inserted (placed under the 1-2nd intercostal space of the thoracotomy incision, in the mid-axillary line)
* having a rigid drainage tube with a diameter of 28-32 Fr
* having a chest tube inserted for the first time.

Exclusion Criteria:

* rib fracture
* pneumonectomy and decortication
* previous thoracic surgery and radiotheraphy
* having a diagnosis of a major neurological problem (as it may affect pain perception and sleep)
* having a diagnosed sleep problem
* a diagnosis of substance or alcohol dependency requiring treatment
* any musculoskeletal problem that prevents positioning in bed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Level | Pain scoring: The first pain scoring was be done on the patient's first day at the clinic before giving the Pleural Irritation Prevention Position at bedtime. The second pain scoring was be done at the first hour when the patient wakes up in the morning
  McGill Pain Questionnaire Short-Form was used for pain assessment. The Verbal Pain Scale, contained in the McGill Pain Questionnaire Short-Form, measured pain intensity at the four-hour mark rating pain of 0 - 5 with 0 = no pain, 1 = mild pain, 2 = discomforting pain, 3 distressing pain, 4 = horrible pain and 5 = excruciating pain.
Sleep quality | Sleep quality: The first sleep quality scoring was be done on the patient's first day of hospitalization, before sleep hour (22:00-23:00 pm). The second measurement was made between 06:00 and 07:00 (am) of the night spent in the Pleural Irritation Preven
  Sleep quality was evaluated with the Richard-Campbell Sleep Questionnaire (RCSQ). Scores between "0-25" indicate very poor sleep quality, and scores between "76-100" indicate very good sleep quality.
Sleep efficiency | Sleep efficiency: Sleep efficiency measurement was made between 06:00 and 07:00 (am) of the night spent in the Pleural Irritation Prevention Position.
  Sleep efficiency during one night's sleep was measured with a polysomniograph device. Sleep efficiency was evaluated between "0-100" and a value between "85-100" was considered effective sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Kol, Professor, Study Chair — Head of Nursing Department
Locations (1):
- Akdeniz University Faculty of Nursing, Antalya, Konyaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study results have not yet been published.

REFERENCES:
- [Background] Charnock Y, Evans D. Nursing management of chest drains: a systematic review. Aust Crit Care. 2001 Nov;14(4):156-60. doi: 10.1016/s1036-7314(05)80058-x. PMID 11806513
- [Background] Lavigne, G. (2007). S15. A Pain perception during sleep. Sleep Medicine, (8), S21.
- [Background] Bastuji, H. (2017). S167 Sensory workup during NONREM sleep. Clinical Neurophysiology, 128(9), e232.
- [Background] Baranwal N, Yu PK, Siegel NS. Sleep physiology, pathophysiology, and sleep hygiene. Prog Cardiovasc Dis. 2023 Mar-Apr;77:59-69. doi: 10.1016/j.pcad.2023.02.005. Epub 2023 Feb 24. PMID 36841492
- [Background] Fox V, Gould D, Davies N, Owen S. Patients' experiences of having an underwater seal chest drain: a replication study. J Clin Nurs. 1999 Nov;8(6):684-92. doi: 10.1046/j.1365-2702.1999.00307.x. PMID 10827615
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509